CLINICAL TRIAL: NCT01554527
Title: Sleep-Disordered Breathing and CPAP After Adenotonsillectomy in Children
Brief Title: Continuous Positive Airway Pressure (CPAP) After Adenotonsillectomy in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Michigan Technological University (Other)
Responsible Party: Principal Investigator, Ronald D. Chervin, M.D., M.S., Professor of Neurology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F029661-00; 1R01HL105999-01A1 (NIH)
Record Dates: First submitted 2012-03-01; First posted 2012-03-15 (Estimated); Results first posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Child Behavior Disorders; Attention Deficit Disorder With Hyperactivity; Disorders of Excessive Somnolence
Keywords: polysomnography; child; continuous positive airway pressure; tonsillectomy; neuropsychological tests; cognition; sleepiness; behavior
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Child Behavior Disorders; Attention Deficit Disorder with Hyperactivity; Disorders of Excessive Somnolence; Sleepiness; Behavior | interventions — Continuous Positive Airway Pressure; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CPAP treatment (Experimental): Children randomized to this arm will receive 6 months of CPAP (or BPAP) treatment, beginning at approximately 4 months after AT, in addition to standard of care. For analysis purposes those children who were non-adherent (CPAP use <4 hours per night) vs. adherent (CPAP use at least 4 hours per night) will be analyzed separately.
  Interventions: Procedure: CPAP treatment
- No CPAP treatment (Other): Children randomized to this comparison arm will not be treated with CPAP or BPAP, but will be followed for approximately 10 months after AT while receiving standard of care.
  Interventions: Other: No CPAP treatment

INTERVENTIONS:
Procedure: CPAP treatment — 6 months of treatment with PAP (CPAP or BPAP)
  Other Names: Continuous positive airway pressure device (CPAP); Bi-level positive airway pressure device (BPAP); Positive Airway Pressure device (PAP)
  Arms: CPAP treatment
Other: No CPAP treatment — Children randomized to the comparison group will receive routine care
  Other Names: Comparison group; Control group
  Arms: No CPAP treatment

SUMMARY:
Obstructive sleep-disordered breathing (SDB) affects 2-3% of children and may lead to problems with nighttime sleep and daytime behavior, learning, sleepiness, and mood. Adenotonsillectomy (AT) is the second most common surgical procedure in children. It is now performed more often for suspected SDB than for any other indication. However, recent studies indicate that many if not most children still have SDB after AT, and many still have learning or behavioral problems associated with SDB. The goals of this study are: (1) to assess the extent that behavior, cognition, and sleepiness in children can improve with Continuous positive airway pressure (CPAP) treatment after AT, and (2) to identify which patients stand to gain most from post-operative assessment and treatment.

DETAILED DESCRIPTION:
Obstructive sleep-disordered breathing (SDB) affects at least 2-3% of children and may have substantial adverse impact on behavior and cognition. Adenotonsillectomy (AT), the second most common surgical procedure in children, is now performed more often for suspected SDB than for any other indication. However, recent studies among an increasingly obese population now show something alarming: many if not most children still have SDB after AT, and many still suffer from residual neurobehavioral morbidity. Furthermore, the investigators' ongoing, 12-year, NIH-funded research has shown that standard preoperative polysomnographic measures of SDB do not consistently predict post-AT improvement in behavior and cognition. This may arise in part because many children after AT still have SDB, and because linear relationships between standard SDB measures and neurobehavioral morbidity may not exist. Even at subtle levels, SDB may promote significant neurobehavioral morbidity. Some have suggested that polysomnography may be more important after AT than before AT. However, in practice few children receive polysomnography before AT, and even fewer after AT, when continuous positive airway pressure (CPAP) could still provide definitive relief from SDB. Preliminary data from our group suggest that CPAP after AT is well-tolerated by most children and may provide significant benefit. However, virtually no published evidence exists to address critical clinical questions: which children benefit most from CPAP after AT; what role can clinical symptoms or polysomnography play in that determination; and what neurobehavioral gains are achieved by CPAP after AT?

The investigators therefore will undertake a highly practical, clinical study with two main goals: (1) to assess the extent that behavior, cognition, and sleepiness in children can improve with CPAP after AT, and (2) to identify which patients stand to gain most from post-operative assessment and treatment. This research will use reversible SDB-related neurobehavioral morbidity as the criteria by which to judge the utility of clinical symptoms and polysomnography in identification of candidates for CPAP after AT.

ELIGIBILITY:
Inclusion Criteria:

1. Children ages 5-12 years old,
2. Scheduled for an adenotonsillectomy for treatment of sleep apnea,
3. Child must provide assent, and
4. Parent or legal guardian must be able to speak and read English, and agree to the study.

Exclusion Criteria:

1. No siblings of children already enrolled in the study,
2. Children who expect to have another surgery (in addition to AT) during the period of participation in this study,
3. Neurological, psychiatric, or medical conditions, or social factors that may affect test results, prevent children from returning for required study visits, or interfere with the study treatment, or
4. Certain medications that affect sleepiness or alertness, for example:

   * Stimulants (such as Ritalin, Adderall, or Concerta),
   * Sleep aides (such as Melatonin, Ambien, or Ativan), or
   * Sedating medicines (such as Benadryl, Klonopin, Xanax, or Valerian).

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2012-03; Primary Completion 2017-10-29 (Actual); Study Completion 2017-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald D. Chervin, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 120 consented, 105 were randomized to CPAP or control. (Of the 15 who weren't randomized, 8 were lost to follow up; the other withdrew for various reasons)
Groups:
- Control Group (Surgery Only - no CPAP): The participants who were not assigned to CPAP
- CPAP After Surgery (Adherent): Those participants assigned to CPAP who had at least 4 hours of electronically recorded CPAP use per night
- CPAP After Surgery (Non-adherent): Those participants assigned CPAP who did not have at least 4 hours of electronically recorded CPAP use per night.
Period: Overall Study
Arm/Group | Control Group (Surgery Only - no CPAP) | CPAP After Surgery (Adherent) | CPAP After Surgery (Non-adherent)
Started | 34 | 38 | 33
Crossed Over to Control | 0 | 0 | 2
Had CPAP Titration | 0 (No control group members received CPAP (definitionally)) | 38 | 30
Initiated CPAP Treatment at Home | 0 | 38 | 28
Completed as a Control | 33 | 0 | 1
Completed | 33 | 38 | 25
Not Completed | 1 | 0 | 8
Not completed — Withdrawal by Subject | 1 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 4
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group (Surgery Only - no CPAP) | CPAP After Surgery (Adherent) | CPAP After Surgery (Non-adherent) | Total
Number analyzed (Participants) | 34 | 38 | 33 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.9 (2.0) | 8.3 (2.2) | 8.0 (2.0) | 8.1 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 21 | 16 | 50
  Male | 21 | 17 | 17 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 0 | 7
  Not Hispanic or Latino | 29 | 36 | 33 | 98
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 5 | 8 | 14
  White | 28 | 29 | 19 | 76
  More than one race | 4 | 3 | 5 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34 | 38 | 33 | 105
Behavioral Index [Mean (Standard Deviation); unit: units on a scale (T-Score)] — Computation of T-scores (mean of 50, SD of 10). Minimum value < 10, maximum value >90, SD=10. Higher scores indicate worse behavior Population: Behavioral Index was not available for one control
  units on a scale (T-Score)
    number analyzed (Participants) | 33 | 38 | 33 | 104
    (all) | 61.6 (13.4) | 56.5 (11.3) | 57.8 (11.6) | 58.5 (12.1)
NIH Toolbox Age adjusted composite score [Mean (Standard Deviation); unit: units on a scale] — Scores are reported as Standardized scores with a mean of 100, and SD of 15. Minimum value 40, maximum value 160. Higher scores are good Population: Subject ages too young for this particular test so their data are not included
  units on a scale
    number analyzed (Participants) | 34 | 38 | 29 | 101
    (all) | 95.7 (11.9) | 96.2 (12.3) | 93.9 (11.6) | 95.1 (11.6)
Epworth Sleepiness Scale [Mean (Standard Deviation); unit: units on a scale] — Modified Epworth for children (Melendres et al 2004); 8 questions with each item summed; minimum score 0, maximum score 24. No SD. Higher scores are worse Population: Epworth sleepiness scale score missing for one participant
  units on a scale
    number analyzed (Participants) | 34 | 37 | 33 | 104
    (all) | 7.2 (4.6) | 6.9 (3.9) | 6.4 (3.0) | 6.8 (3.9)
Multiple Sleep Latency Test (MSLT) [Mean (Standard Deviation); unit: minutes] — Mean sleep latency of five 30-min nap attempts. Minimum would be 0 and maximum would be 30 (average of all naps). Shorter times indicate higher sleepiness.
  minutes | 24.7 (6.0) | 25.9 (4.6) | 24.4 (5.4) | 25.0 (5.3)
Quality of Life [Mean (Standard Deviation); unit: units on a scale] — Quality of Life is measured by the PedsQL on a scale of 0 to 100, with higher scores meaning better quality of life
  units on a scale | 78.2 (13.7) | 78.7 (16) | 77.3 (17.2) | 78.1 (14.9)
Academic Achievement Score [Mean (Standard Deviation); unit: units on a scale] — Scores are reported as Standardized scores with a mean of 100 and SD of 15. Minimum value 40; Maximum value 160. Higher scores are better
  units on a scale | 104.1 (13.4) | 107.2 (14.6) | 102.1 (10.7) | 104.6 (13.1)
Fluid Cognition Composite Age Adjusted score [Mean (Standard Deviation); unit: units on a scale] — Scores are reported as Standardized scores with a mean of 100 and SD of 15. Minimum value 40; Maximum value 160; SD = 15; higher scores are better Population: Subject age was too young for this particular test, so their data is not included.
  units on a scale
    number analyzed (Participants) | 34 | 38 | 30 | 102
    (all) | 97.3 (13.2) | 96 (14.2) | 93.9 (11.6) | 95.8 (13.1)
(Apnea-Hypopnea Index (AHI) [Mean (Standard Deviation); unit: events/hour] | 2.4 (2.0) | 2.2 (1.7) | 2.1 (2.0) | 2.2 (1.9)
Sleep Related Breathing Disturbances (SBRD) sub-scale of Pediatric Sleep Questionnaire [Mean (Standard Deviation); unit: Ratio] — The ratio of number of positive responses to the questionnaire divided by the total number of responses. Minimum 0 maximum 1. A ratio of 0.33 or more suggests high risk for sleep-disordered breathing.
  Ratio | 0.36 (0.24) | 0.32 (0.21) | 0.37 (0.17) | 0.35 (0.21)

OUTCOME MEASURES:

1. Primary Outcome: Change in Behavioral Index After 6 Months of CPAP or No-CPAP
Description: The sum of the T-scores of The Conners' Parent Rating Scales (CPRS-R:L, ADHD index) and the Child Behavior Checklist (CBCL, Attention Deficit/Hyperactivity Problems) are used to construct the primary study outcome measure Behavioral Index. Behavioral index is a T score (adjusted for age and gender) with a range of "<10" to ">90" - where higher scores mean worse behavior and lower scores mean better behavior, so a negative change score represents an improvement in behavior. T-scores with a mean of 50 and SD of 10 are computed.
Time Frame: assessed as change from baseline to 6 months of CPAP therapy or no-CPAP
Population: Data for two participants in the control group are not available.
Measure: Mean (Standard Deviation); unit: T score
Groups:
- CPAP After Surgery (Non-adherent): Those participants assigned CPAP who did not have at least 4 hours of electronically recorded CPAP use per night over the last 60 days of the 6 month usage period
- CPAP After Surgery (Adherent): Those participants assigned to CPAP who had an average of at least 4 hours of electronically recorded CPAP use per night over the last 60 days of the 6 month usage period
Arm/Group | Control Group (Surgery Only - no CPAP) | CPAP After Surgery (Non-adherent) | CPAP After Surgery (Adherent)
Number analyzed (Participants) | 32 | 25 | 38
T score | -2.7 (5.8) | .9 (4.8) | -1.2 (6.3)
Statistical Analysis 1: Comparison: Control Group (Surgery Only - no CPAP) vs CPAP After Surgery (Non-adherent) vs CPAP After Surgery (Adherent); Intent to treat for controls vs. treatment (adherent/non-adherent); Test type: Superiority; p = 0.07, t-test, 2 sided

2. Secondary Outcome: Change in Cognition as Shown by NIH Toolbox Composite Score
Description: Scores are reported as standardized scores with a mean of 100 and SD of 15. Minimum value 40 and Maximum value 160. Higher scores are better
Time Frame: assessed as change from baseline to 6 months of CPAP therapy or no-CPAP
Population: Lower numbers of participants analyzed are shown here because the tool is not appropriate for younger children
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group (Surgery Only - no CPAP) | CPAP After Surgery (Non-adherent) | CPAP After Surgery (Adherent)
Number analyzed (Participants) | 27 | 23 | 38
score on a scale | 5.5 (9.5) | 2.8 (9.8) | 3.9 (7.8)
Statistical Analysis 1: Comparison: Control Group (Surgery Only - no CPAP) vs CPAP After Surgery (Non-adherent) vs CPAP After Surgery (Adherent); Intent to treat for controls vs. treatment (adherent/non-adherent); Test type: Superiority; p = 0.34, t-test, 2 sided

3. Secondary Outcome: Change in Sleepiness as Measured by Epworth Sleepiness Scale
Description: Epworth Sleepiness Scale scores range from 0 to 24 where higher scores mean greater sleepiness.
Time Frame: assessed as change from baseline to 6 months of CPAP therapy or no-CPAP
Population: Data for two participants are not available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group (Surgery Only - no CPAP) | CPAP After Surgery (Non-adherent) | CPAP After Surgery (Adherent)
Number analyzed (Participants) | 33 | 25 | 37
score on a scale | -1.6 (3.7) | -1.0 (2.2) | -1.9 (3.8)
Statistical Analysis 1: Comparison: Control Group (Surgery Only - no CPAP) vs CPAP After Surgery (Non-adherent) vs CPAP After Surgery (Adherent); Intent to treat for controls vs. treatment (adherent/non-adherent); Test type: Superiority; p = 0.93, t-test, 2 sided

4. Secondary Outcome: Change in Sleepiness After AT as Measured by Multiple Sleep Latency Test (MSLT)
Description: Multiple Sleep Latency Test (MSLT) is an objective measure of sleepiness determined by measure of brain waves and other physiological signals over a 30 minute period. This is measured for five 30 minute periods across the day and average latency to sleep for each participant across those times were used to calculate the mean sleep latency. The score is measured in how quickly one would fall asleep, measured in minutes, so a negative number of minutes in the change score means that participants fell asleep more quickly than previously.
Time Frame: assessed as change from baseline to 6 months of CPAP therapy or no-CPAP
Population: Data for one participant are not available
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control Group (Surgery Only - no CPAP) | CPAP After Surgery (Non-adherent) | CPAP After Surgery (Adherent)
Number analyzed (Participants) | 33 | 25 | 38
minutes | -1.8 (4) | -1.3 (5.1) | -1.1 (4.3)
Statistical Analysis 1: Comparison: Control Group (Surgery Only - no CPAP) vs CPAP After Surgery (Non-adherent) vs CPAP After Surgery (Adherent); Intent to treat for controls vs. treatment (adherent/non-adherent); Test type: Superiority; p = 0.5, t-test, 2 sided

5. Secondary Outcome: Change in Quality of Life as Measured by Peds QL
Description: Peds-QL is a quality of life symptom measurement with a score range of 0 to 100. Higher scores are better quality of life
Time Frame: assessed as change from baseline to 6 months of CPAP therapy or no-CPAP
Population: Data for one participant is not available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group (Surgery Only - no CPAP) | CPAP After Surgery (Non-adherent) | CPAP After Surgery (Adherent)
Number analyzed (Participants) | 33 | 25 | 38
score on a scale | 4.1 (9.0) | 0.5 (10.2) | 2.4 (12.1)
Statistical Analysis 1: Comparison: Control Group (Surgery Only - no CPAP) vs CPAP After Surgery (Non-adherent) vs CPAP After Surgery (Adherent); Intent to treat for controls vs. treatment (adherent/non-adherent); Test type: Superiority; p = 0.25, t-test, 2 sided

6. Secondary Outcome: CPAP Adherence as Measured by Number of Participants Who Used the CPAP Consistently.
Description: CPAP adherence data will be downloaded from CPAP machines. It is defined for this study as using the CPAP machine for at least an average of 4 hours per night during the last 60 days of the assignment.
Time Frame: Starting at 4 months after AT and continuing through 10 months after AT
Measure: Count of Participants; unit: Participants
Groups:
- CPAP Group: Participants who were assigned to CPAP use.
Arm/Group | CPAP Group
Number analyzed (Participants) | 71
Participants | 38

7. Other Pre Specified Outcome: Change in Cognition as Measured by Fluid Cognition Scores
Description: Scores are reported as standardized scores with a mean of 100 and SD of 15. Minimum value 40, Maximum value 160. Higher scores are better
Time Frame: assessed as change from baseline to 6 months of CPAP therapy or no-CPAP
Population: Lower numbers are shown here as the tool is not appropriate for younger children
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group (Surgery Only - no CPAP) | CPAP After Surgery (Non-adherent) | CPAP After Surgery (Adherent)
Number analyzed (Participants) | 29 | 23 | 38
score on a scale | 6.7 (12.4) | 1.7 (11.5) | 3.4 (10.1)

8. Other Pre Specified Outcome: Change in Cognition After AT as Shown by Academic Achievement
Description: Academic achievement mean score is a standardized score with a mean of 100 and SD 15. Minimum value 40 and Maximum value 160. Higher scores are better
Time Frame: assessed as change from baseline to 6 months of CPAP therapy or no-CPAP
Population: Data from two participants are not available
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group (Surgery Only - no CPAP) | CPAP After Surgery (Non-adherent) | CPAP After Surgery (Adherent)
Number analyzed (Participants) | 32 | 25 | 37
units on a scale | -1.0 (5.6) | 1.1 (4.7) | -2.5 (8.6)

ADVERSE EVENTS:
Time Frame: Adverse events were followed from consent (which could be before surgery or after surgery) until 10 months after surgery equating to six months after assignment.
Description: Based on the adverse event collection structure, it bears noting that some reported AEs may have happened prior to assignment to CPAP or no CPAP use, to participants who ended up reaching baseline visit (4 months after surgery). Since both adherent and non-adherent CPAP participants received CPAP with minimum 1 night of CPAP, these 2 groups were combined for the purposes of AE reporting in order to determine whether any CPAP exposure vs control group (no CPAP) had a different proportion of AE's.
Groups:
- CPAP Treatment Group on CPAP: Children randomized to this arm were assigned and began up to 6 months of CPAP treatment, beginning at approximately 4 months after AT, in addition to standard of care. This arm shows AEs that happened to participants randomized to CPAP but who didn't cross over to the No CPAP group prior to sleep lab. (n=69; original n=71 minus n=2 who crossed over to no-CPAP group). Since both adherent and non-adherent CPAP participants received CPAP and had at minimum one night of CPAP exposure, these two groups were combined for the purposes of AE reporting in order to determine whether any CPAP exposure vs control group (no CPAP) had a different proportion of AE's.
- No CPAP Treatment Group: Children shown in this comparison arm were randomized to NO CPAP or were crossed over to No CPAP prior to any CPAP use or CPAP trial in sleep lab.) (N = 36, original 34 plus two crossed over from those randomized to CPAP)
- Non-randomized Participants: Participants who were consented but withdrew prior to randomization (n = 15)
Arm/Group | CPAP Treatment Group on CPAP | No CPAP Treatment Group | Non-randomized Participants
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/36 | 0/15
Serious Adverse Events (participants affected / at risk) | 6/69 | 7/36 | 4/15
Other Adverse Events (participants affected / at risk) | 59/69 | 26/36 | 7/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CPAP Treatment Group on CPAP (N=69) | No CPAP Treatment Group (N=36) | Non-randomized Participants (N=15)
Hospitalization for ashthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Post-operative hospitalization (Surgical and medical procedures) | 4 | 7 | 4 — Pre-scheduled hospitalizations or within 48 hours of surgery (prior to randomization in the trial)
ER admission due to panic attack (Psychiatric disorders) | 1 | 0 | 0 — This occurred after signing consent but prior to randomization
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CPAP Treatment Group on CPAP (N=69) | No CPAP Treatment Group (N=36) | Non-randomized Participants (N=15)
Allergic Reaction (Immune system disorders) | 8 | 5 | 0
Anxiety (Psychiatric disorders) | 12 | 8 | 0
Asthma Exacerbation (Respiratory, thoracic and mediastinal disorders) | 17 | 5 | 0
Behavior Issues (Social circumstances) | 11 | 4 | 0
Cold Symptoms (General disorders) | 38 | 16 | 2
Constipation (Gastrointestinal disorders) | 4 | 0 | 0
Ear Pain (Ear and labyrinth disorders) | 2 | 0 | 2
Enuresis (Renal and urinary disorders) | 5 | 0 | 0
Flu-like Symptoms (General disorders) | 0 | 3 | 0
GI Distress (Gastrointestinal disorders) | 7 | 1 | 1
Headache (Nervous system disorders) | 3 | 2 | 0
HFMD (Infections and infestations) | 0 | 2 | 0
Life Event or Change (Social circumstances) | 2 | 5 | 1
Molluscum Contagiosum (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Pink Eye (Eye disorders) | 2 | 2 | 0
Skin Irritation (Skin and subcutaneous tissue disorders) | 42 | 12 | 0
Stomach Flu (Gastrointestinal disorders) | 14 | 5 | 0
Strep Throat (Infections and infestations) | 1 | 1 | 1
Unrelated Accident (Injury, poisoning and procedural complications) | 22 | 9 | 1
Upper Respiratory Infection (Infections and infestations) | 7 | 6 | 2
Voice Alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Vomiting (Gastrointestinal disorders) | 7 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT01554527/Prot_SAP_000.pdf